CLINICAL TRIAL: NCT05796635
Title: An Investigation Into the Efficacy of Herpecin L at Reducing the Frequency and Severity of Cold Sores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Focus Consumer Healthcare (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20274
Record Dates: First submitted 2023-03-09; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-04

CONDITIONS: Cold Sores
MeSH Terms: conditions — Herpes Labialis | interventions — Allantoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herpecin L (Experimental): Participants will use Herpecin L Everyday Protection lip balm.
  Interventions: Other: Herpecin L
- Controlled Arm (No Intervention): Participants will not use any cold sore products or lip balms.

INTERVENTIONS:
Other: Herpecin L — Participants in the Herpecin L arm will use the test product daily as a preventive product by applying the product twice daily. Also, participants will be told they can reapply the product if going outside into the cold, wind, or sun. If participants in the Herpecin L arm do experience a cold sore or fever blister, they will be instructed to use the product at the first sign of the cold sore and then at least four more times during the day until the cold sore is gone (they can use the product more often if they plan to go outside into the cold, sun, or wind).
  Arms: Herpecin L

SUMMARY:
Focus Consumer Healthcare has developed Herpecin L. Herpecin L combines many different ingredients hypothesized to promote quick healing and symptom reduction from cold sores.

ELIGIBILITY:
Inclusion Criteria:

* Male Female between 18-60 years of age.
* Must be in good health with no significant chronic conditions and a BMI under 35.
* Must experience regular cold sores or fever blisters
* Must agree to avoid daily lip balm or another product designed to alleviate their cold sore (e.g., Abreva or other over-the-counter cold sore products).

Exclusion Criteria:

* Suffers from pre-existing conditions that would prevent them from adhering to the protocol including chronic conditions such as oncological or psychiatric disorders.
* Anyone with known severe allergic reactions.
* Unwilling to follow the study protocol.
* Currently pregnant, breastfeeding, or wanting to become pregnant for the duration of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
The primary aim of this research is to understand the changes in cold sore severity. | 12 weeks
  Cold sore severity will be measured via survey and cold sore severity grading. Symptom severity is rated on a scale of 0 (Not a problem) to 6 (Severe)

SECONDARY OUTCOMES:
The secondary objective of this trial is to examine differences in cold sore frequency between the two groups. | 12 weeks
  Cold sore frequency will be measured via a self-reported survey measuring the frequency of cold sore occurrence during the study period compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States